CLINICAL TRIAL: NCT04650230
Title: High Flow Nasal Cannula Therapy (HFNC) Versus Nasal Positive Airway Pressure and or Nasal Positive Pressure Ventilation (NCPAP/ NPPV) in Infants With Severe Bronchiolitis
Brief Title: HFNC Versus NCPAP/ NPPV in Infants With Severe Bronchiolitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Tunis (Other)
Responsible Party: Principal Investigator, Aida Borgi, Professor, Children's Hospital of Tunis
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: RPP1
Record Dates: First submitted 2020-11-25; First posted 2020-12-02 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Bronchiolitis
MeSH Terms: conditions — Bronchiolitis | interventions — Continuous Positive Airway Pressure; Equipment and Supplies

ARMS (2):
- high flow nasal cannula (HFNC) (Active Comparator): Participants in the HFNC group received heated and humidified gas flow with the Fisher & Paykel Healthcare HFNC system. The flow rate was usually started at the maximum flow rate for the size of cannula and a constant flow temperature of 37 °C.The flow rate will be progressively decreased when inspired fraction of oxygen (FiO2) was inferior to 30 percent (%).
  Interventions: Device: nasal continuous positive airway pressure / nasal positive pressure ventilation (NCPAP/NPPV) and high flow nasal cannula (HFNC) devices
- nasal continuous positive airway pressure / nasal positive pressure ventilation (NCPAP/NPPV) (Active Comparator): Participants in the CPAP/NPPV group received for first CPAP using a neonatal ventilator. The recommended starting pressure for CPAP was +6 centimeter of water (cmH2O). Positive continuous pressure could be increased to a maximum of +8 cmH2O. Optimal positive end expiratory pressure (PEEP) was what could maintain SpO2 at 94 per cent using the lowest fraction of inspired oxygen. PEEP will be decreased progressively of 1cmH2O every 6 hours from the optimal PEEP when FiO2 was inferior to 30% and there is no increase of work of breath.
  Interventions: Device: nasal continuous positive airway pressure / nasal positive pressure ventilation (NCPAP/NPPV) and high flow nasal cannula (HFNC) devices

INTERVENTIONS:
Device: nasal continuous positive airway pressure / nasal positive pressure ventilation (NCPAP/NPPV) and high flow nasal cannula (HFNC) devices

SUMMARY:
The purpose of the study was to test the null hypothesis that there is no difference between nasal continuous positive airway pressure / nasal positive pressure ventilation (NCPAP/NPPV) and high flow nasal cannula (HFNC) devices when applied as a first non-invasive respiratory support mode for severe bronchiolitis

DETAILED DESCRIPTION:
The authors conducted a randomized controlled trial in the PICU of Children's hospital of Tunis. Participants aged from 7 days to 6 months, were eligible if all inclusion criteria were verified.

On admission, demographic and clinical data were collected. When a participant met the inclusion criteria, respiratory support was randomly allocated as high flow nasal cannula (HFNC) or nasal continuous positive airway pressure / nasal positive pressure ventilation (CPAP/NPPV).

Clinical parameters were monitored at treatment start and every 6 hours during the first 24 hours and then twice daily thereafter.

Participants in the HFNC group received heated and humidified gas flow with the Fisher & Paykel Healthcare HFNC system. The flow rate was usually started at the maximum flow rate for the size of cannula and a constant flow temperature of 37 °C.The flow rate will be progressively decreased when inspired fraction of oxygen (FiO2) was inferior to 30 percent (%).

Participants in the CPAP/NPPV group received for first CPAP using a neonatal ventilator. The recommended starting pressure for CPAP was +6 centimeter of water (cmH2O). Positive continuous pressure could be increased to a maximum of +8 cmH2O. Optimal positive end expiratory pressure (PEEP) was what could maintain SpO2 at 94 per cent using the lowest fraction of inspired oxygen. PEEP will be decreased progressively of 1cmH2O every 6 hours from the optimal PEEP when FiO2 was inferior to 30% and there is no increased work of breathing.

If CPAP failed to improve clinical respiratory distress, infant was allocated to NPPV strategy. Clinicians were not be authorized to change from CPAP to HFNC but if HFNC failed, they had to change HFNC to CPAP/NPPV strategy ventilation before intubation.

Treatment failure criteria were urgent need to intubation or FiO2 superior to 60 % to maintain SpO2 ≥ 90% or increased work of breathing.

Sample size (134 per group) was calculated on the basis of Type I error equal to 0,05, on statistical power equal to 0.95 on failure rate among controls estimated at 30% and assuming a minimum difference of failure rate to declare the superiority of intervention equal to 20%. A dropout rate equal to 20% was used for this calculation.

Statistical Analysis Comparison of proportions was performed using Fisher exact test, and Student t test was used for comparison of means. For all analyses, significance level was defined as p < 0.05.

All statistical analyses were performed using Microsoft Excel 365.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of bronchiolitis defined as the first viral episode of respiratory distress before 2 years of aging, presenting with rhinitis, tachypnea, cough, wheezing, prolonged expiratory time, crackles and use of accessory muscles, with or without fever, with or without infiltrate on the chest X ray
* bronchiolitis severity Wang modified score ≥ 10

Exclusion Criteria:

* recurrent wheezing
* heart disease
* chronic lung disease
* neuromuscular disease
* primary diagnosis was not bronchiolitis (pneumonia, pertussis)
* critically ill infants who had an immediate need of intubation

Ages: 7 Days to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 268 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Number of participants with HFNC success | during hospitalization, approximatly 6 days
  success was defined by no need of another respiratory support device
Number of participants with CPAP/NPPV success | during hospitalization, approximatly 6 days
  success was defined by no need of another support device

SECONDARY OUTCOMES:
rate of intubation | during hospitalization, approximatly 6 days
  need of intubation

IPD SHARING:
Plan to Share IPD: No